CLINICAL TRIAL: NCT00498862
Title: Catecholamines Can Attenuate Intermittent Hypoxia-Induced Expression of TNF in Human Monocytes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561709069
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2006-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Specific aim To examine the effect of catecholamines on the modulation of intermittent hypoxia induced TNF- in human monocytes from both healthy subjects and OSA patients (2). To map the signaling pathway of catecholamines regulating the intermittent hypoxia induced TNF- expression.

(3). To explore the potential therapeutic effects of  or  agonists/antagonists on intermittent hypoxia induced TNF- expression

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common disease, which occurs in 4% middle-aged men and 2% middle-aged women. The characteristic of OSA is recurrent collapse of upper airway during sleep, which results in intermittent hypoxia and sympathetic activation. Cardiovascular complications associated with OSA include artherosclerosis, hypertension, coronary artery disease and congestive heart failure. Several inflammatory mediators including C-reactive protein (CRP), oxidative stress, adhesion molecules, vascular endothelial growth factor and proinflammatory cytokines, were found to be elevated in OSA, which attribute the developments of cardiovascular diseases in OSA. Our data showed serum levels of TNF were higher in OSA patients than in control subjects. And serum levels of TNF were inversely correlated with the lowest pulse oxygen saturation. After one-month CPAP treatment, serum of TNF could significantly go down. This finding suggested TNF was a good biomarker in studying OSA associated cardiovascular complications.

The presentations of sympathetic hyperactivity in OSA include hypercatecholaminemia and elevated sympathetic tone of peripheral nerve. Hypercatecholaminemia is known for attributing to the development of cardiovascular diseases. Our data showed plasma levels of both epinephrine and norepinephrine were higher in OSA patients than in control subjects. And the elevated catecholamine could go down after one-month CPAP treatment. Meanwhile, our data also showed the plasma levels of catecholamine were highly correlated with serum levels of TNF.

In vivo studies showed both epinephrine and norepinephrine could potentiate LPS-induced expression of TNF through 2 adrenergic receptors. However, the effect of catecholamine on TNF production in human monocytes in the hypoxic microenvironment has never been studied. Our preliminary data showed epinephrine had no effect on TNF expression in human monocyte cell line U937 under normoxic condition but could attenuate the TNF expression under hypoxic condition. Therefore, we hypothesize that catecholamines can modulate intermittent hypoxia induced TNF and further affect the developments of cardiovascular complications in OSA. In this project, we'll use peripheral blood monocytes from healthy subjects and OSA patients as the target cells, which were serially treated with catecholamine  or b antagonists in both normoxic and hypoxic microenvironments, to achieve the following 3 objectives:

1. . To examine the effect of catecholamines on the modulation of intermittent hypoxia induced TNF- in human monocytes from both healthy subjects and OSA patients
2. . To map the signaling pathway of catecholamines regulating the intermittent hypoxia induced TNF- expression.
3. . To explore the potential therapeutic effects of  or  agonists/antagonists on intermittent hypoxia induced TNF- expression

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Peiln Lee, M.D., Principal Investigator — National Taiwan Univerisity Hospital; Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan